CLINICAL TRIAL: NCT00680225
Title: Ranibizumab as Adjuvant Therapy for the Treatment of Choroidal Melanoma
Brief Title: Lucentis as an Adjuvant Therapy With TTT-ICG Based in Choroidal Melanoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: New England Retina Associates (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FVF4290s; NCT00541528 (obsolete NCT alias)
Record Dates: First submitted 2008-05-15; First posted 2008-05-20 (Estimated); Results first posted 2017-04-12 (Actual); Last update posted 2017-04-12 (Actual); Status verified 2017-04

CONDITIONS: Choroidal Melanoma
Keywords: Choroidal melanoma; Lucentis; TTT-ICG
MeSH Terms: conditions — Uveal Melanoma | interventions — Ranibizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lucentis Injection (Experimental): Intravitreal injection of ranibizumab (0.5mg) once a month for 6 months and transpupillary thermotherapy enhanced with Indocyanine Green (ICG) dye, once or twice starting at 2nd month.
  Interventions: Drug: Ranibizumab injection and TTT - ICG based

INTERVENTIONS:
Drug: Ranibizumab injection and TTT - ICG based — Intravitreal injection of ranibizumab (0.5mg) once a month for 6 months and transpupillary thermotherapy enhanced with Indocyanine Green (ICG) dye, once or twice starting at 2nd month.
  Other Names: Lucentis injection

SUMMARY:
To report preliminary results on safety and tolerability of intravitreal injection of Ranibizumab (Lucentis) combined with Transpupillary Thermotherapy (TTT)+ Indocyanine Green (ICG)-based photodynamic therapy (PDT) in the treatment of choroidal melanoma.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 yo.
* Primary pigmented or amelanotic choroidal melanoma measurement of 16 mm or less in the largest vessel diameter and 6 mm or less in the apical height.
* Location of the tumor posterior to the equator.
* Documented growth by A/B scan.
* Risk factor for metastasis (thickness greater than 2 mm, symptoms, tumor margin at the optic disc)
* Ability to provide inform consent.
* Comply with the study assessment for the cooperation of the study.

Exclusion Criteria:

* Pregnancy or lactation.
* Premenopausal women not using adequate contraception; surgical sterilization or use of oral contraception, barrier contraception with either a condom or diaphragm or in conjunction with spermicidal gel, an IUD or contraceptive hormon implant or patch.
* Current infection or inflammation in either eye.
* Extension of tumor into the orbit.
* Retinal spread or metastatic disease.
* Any other condition that the investigator believes would pose a significant hazard to the subject if the investigational therapy were initiated.
* Any known allergy to any of the components to be used in the study.
* Participation in another simultaneous medical investigation or trial.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2007-09; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- New England Retina Associates, Hamden, Connecticut, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Lucentis Injection
Started | 10
Completed | 8
Not Completed | 2

BASELINE CHARACTERISTICS:
Population: Baseline Data available for 8 participants
Arm/Group | Lucentis Injection
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 4

OUTCOME MEASURES:

1. Primary Outcome: Mean Tumor Thickness
Time Frame: 12 mo
Measure: Mean (Full Range); unit: mm
Arm/Group | Lucentis Injection
Number analyzed (Participants) | 8
mm | 2.91 [2.5 to 3.5]

2. Secondary Outcome: Visual Acuity Changes
Time Frame: 12 mo
Population: PI has left the institution and summary data are not available.
Arm/Group | Lucentis Injection
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Description: Adverse event data are not available to be reported because the PI left the institution and adverse event data in the required format is unavailable.
Arm/Group | Lucentis Injection
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No